CLINICAL TRIAL: NCT03344289
Title: Linked Color Imaging Versus High-definition White Light Endoscopy for the Detection of Polyps in Patients With Lynch Syndrome. An International, Multicenter, Parallel Randomized Controlled Trial.
Brief Title: Linked Color Imaging Versus High-definition White Light Endoscopy for the Detection of Polyps in Patients With Lynch Syndrome (LCI-LYNCH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: FUJIFILM Europe GmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Prof. Evelien Dekker, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL59002.018.16
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Lynch Syndrome; Colonoscopy
Keywords: Linked-color-imaging; Advanced Imaging Techniques
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: An international, multicenter, parallel randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linked color imaging (Experimental): When the patient is randomized for LCI, the imaging mode is switched to LCI and colonoscopic inspection will take place during withdrawal of the endoscope
  Interventions: Diagnostic Test: Colonoscopy
- High definition white light (Active Comparator): When the patient is randomized for HD-WLE, the imaging mode is switched to HD-WLE and colonoscopic inspection will take place during withdrawal of the endoscope.
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Participants will be randomized towards colonoscopy withdrawal with either LCI or HD-WLE

SUMMARY:
The aim of the present study is to compare polyp detection rates of LCI with high-definition white light endoscopy (HD-WLE) in patients with Lynch syndrome in a parallel, international, multicenter, randomized controlled colonoscopy trial

DETAILED DESCRIPTION:
Rationale: Linked Color Imaging is a push-button endoscopic imaging technique developed to enhance the visibility of the vasculature and architecture of the mucosal surface by narrowing the spectrum of absorbed light. Compared to High-Definition White Light Endoscopy, mucosal surface patterns are better visualized and this could potentially increase the detection of polyps by improving the visibility of colorectal polyps. Patients with Lynch syndrome have accelerated carcinogenesis and even the smallest polyps have malignant potential. Increasing polyp detection rates with new imaging techniques is therefore of importance.

Objective: To compare polyp detection rates of Linked Color Imaging with High-Definition White Light Endoscopy during surveillance colonoscopy in Lynch patients Study design: international, multicentre, parallel, randomized controlled trial Inclusion criteria: Patients diagnosed with Lynch syndrome (proven germline mutation in one of the following MMR genes: MLH1, MSH2, MSH6 or PMS2) aged ≥ 18 years old undergoing surveillance colonoscopy Exclusion criteria: Patients who underwent recent surveillance colonoscopy within 1 year from current exam (e.g. after piecemeal EMR) or patients referred for endoscopic evaluation of known colorectal neoplasia. Patients in whom the colonoscopy is planned for the evaluation of symptoms like rectal blood loss, recent change in bowel habits, weight loss or anemia. Patients with a concurrent diagnosis of (serrated) polyposis syndrome or inflammatory bowel disease. Patients who are unwilling or unable to give informed consent.

Intervention: Included patients will undergo surveillance colonoscopy with either Linked Color Imaging colonoscopy or High-Definition White Light Endoscopy after 1:1 randomization.

Main study parameters/endpoints: Polyp detection rate of Linked Color Imaging versus High-Definition White Light Endoscopy Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Each colonoscopy is associated with a small, but not negligible risk of bleeding (~1.5%) or perforation (~0.1%). The use of LCI does not increase the risk of endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lynch-syndrome, with a germline mutation in one of the MMR genes (MLH1, MSH2, MSH6, PMS2)
* Age >18 years
* Surveillance colonoscopy for Lynch syndrome.

Exclusion Criteria:

* Recent surveillance colonoscopy within 1 year from current exam (e.g. after piecemeal EMR) or patients referred for endoscopic evaluation of known colorectal neoplasia.
* Colonoscopy planned for the evaluation of symptoms like rectal blood loss, recent change in bowel habits, weight loss or anemia.
* Patients with a concurrent diagnosis of (serrated) polyposis syndrome or inflammatory bowel disease.
* Patients who are unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2018-01-21 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
polyp detection rates | 2 years
  The aim of the present study is to compare polyp detection rates of LCI with high-definition white light endoscopy (HD-WLE) in patients with Lynch syndrome in a parallel, international, multicenter, randomized controlled colonoscopy trial.

SECONDARY OUTCOMES:
mean number of detected polyps | 2 years
adenoma detection rate | 2 years
mean number of adenomas | 2 years
mean number of serrated polyps | 2 years
mean duration of procedures | 2 years
sensitivity, specificity, and accuracy of optical diagnosis on a per polyp basis | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Houwen BBSL, Hazewinkel Y, Pellise M, Rivero-Sanchez L, Balaguer F, Bisschops R, Tejpar S, Repici A, Ramsoekh D, Jacobs MAJM, Schreuder RM, Kaminski MF, Rupinska M, Bhandari P, van Oijen MGH, Koens L, Bastiaansen BAJ, Tytgat KM, Fockens P, Vleugels JLA, Dekker E. Linked Colour imaging for the detection of polyps in patients with Lynch syndrome: a multicentre, parallel randomised controlled trial. Gut. 2022 Mar;71(3):553-560. doi: 10.1136/gutjnl-2020-323132. Epub 2021 Mar 18. PMID 34086597